CLINICAL TRIAL: NCT04914936
Title: A Phase 1, Single-Center, Open-Label, Fixed-Sequence, 2-Period, 3-Part Study to Evaluate the One-Way Interaction of Calcium Carbonate, Omeprazole, or Rifampin on ACP-196 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the One-way Interaction of Calcium Carbonate, Omeprazole, or Rifampin on ACP-196
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-HV-004
Record Dates: First submitted 2021-05-21; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Healthy Participants
Keywords: Acalabrutinib; ACP-196; Healthy participants; Pharmacokinetics; PK; Safety
MeSH Terms: interventions — acalabrutinib; Calcium Carbonate; Omeprazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: ACP-196 and Calcium carbonate (Experimental): Participants will receive a single oral dose of ACP-196 100 mg capsule on Day 1 of Period 1 and a single oral dose of calcium carbonate 1 g tablet coadministered with a single oral dose of ACP-196 100 mg capsule on Day 1 of Period 2.
  Interventions: Drug: ACP-196; Drug: Calcium carbonate
- Part 2: ACP-196 and Omeprazole (Experimental): Participants will receive a single oral dose of ACP-196 100 mg capsule on Day 1 of Period 1 and oral dose of omeprazole 40 mg capsules once daily (QD) for 5 consecutive days coadministered with a single oral dose of ACP-196 100 mg capsule on Day 5 of Period 2.
  Interventions: Drug: ACP-196; Drug: Omeprazole
- Part 3: ACP-196 and Rifampin (Experimental): Participants will receive a single oral dose of ACP-196 100 mg capsule on Day 1 of Period 1 and oral dose of rifampin 600 mg capsule QD for 9 consecutive days coadministered with a single oral dose of ACP-196 100 mg capsule on Day 1 and Day 9 of Period 2.
  Interventions: Drug: ACP-196; Drug: Rifampin

INTERVENTIONS:
Drug: ACP-196 — Participants will receive a single oral dose of ACP-196 100 mg capsule on Day 1 of Period 1 in Part 1, Part 2, and Part 3; and on Day 1 of Period 2 in Part 1, Day 5 of Period 2 in Part 2, and Day 1 and Day 9 of Period 2 in Part 3.
  Other Names: Acalabrutinib
Drug: Calcium carbonate — Participants will receive a single oral dose of calcium carbonate 1 g tablet on Day 1 of Period 2 in Part 1.
  Arms: Part 1: ACP-196 and Calcium carbonate
Drug: Omeprazole — Participants will receive multiple oral doses of omeprazole 40 mg capsules QD for 5 consecutive days in Period 2 of Part 2.
  Arms: Part 2: ACP-196 and Omeprazole
Drug: Rifampin — Participants will receive multiple oral doses of rifampin 600 mg capsule QD for 9 consecutive days in Period 2 of Part 3.
  Arms: Part 3: ACP-196 and Rifampin

SUMMARY:
The study will evaluate one-way interaction of calcium carbonate, omeprazole, or rifampin on ACP-196.

DETAILED DESCRIPTION:
This is a 3-part study. Each part will be conducted as an open-label, 2-period, fixed-sequence study. All the study parts will be conducted concurrently and the participants will receive the study treatment in all the parts after an overnight fast. In each part, 24 healthy, non-tobacco using, men and women will be enrolled, to ensure 22 participants complete each part. Each participant will participate in only one study part. In Part 1, a single oral dose of ACP-196 100 mg capsule will be administered on Day 1 of Period 1 (Treatment A), and a single oral dose of calcium carbonate 1 g tablets will be coadministered with a single oral dose of ACP-196 100 mg on Day 1 of Period 2 (Treatment B). In Part 2, a single oral dose of ACP-196 100 mg capsule will be administered on Day 1 pf Period 1 (Treatment C) and oral doses of omeprazole 40 mg capsules once daily (QD) for 5 consecutive days with a single oral dose of ACP-196 100 mg capsule coadministered on Day 5 of Period 2 (Treatment D). In Part 3, a single oral dose of ACP-196 will be administered on Day 1 of Period 1 (Treatment E) and oral dose of rifampin 600 mg capsule QD for 9 consecutive days with a single oral dose of ACP-196 100 mg capsule coadministered on Day 1 and Day 9. Participants will be screened within 28 days before the dose. There will be no washout between the dose in Period 1 and the first dose in Period 2. Participants will be contacted approximately 14 days after the last dose of study drug for adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dose.
* Body mass index (BMI) >= 18.0 and =< 32.0 kg/m^2 at screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or electrocardiograms (ECGs), as deemed by the principal investigator (PI). Liver function tests must be =< upper limit of normal range (ULN).
* Women must be of non-childbearing status and must have negative serum pregnancy test results.
* Men of reproductive potential to follow protocol defined contraception methods.
* Able to swallow multiple capsules.

Exclusion Criteria:

* Participant is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI.
* History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* Presence of any clinically significant, ongoing systemic bacterial, fungal, or viral infections in the opinion of the PI.
* History or presence of alcoholism or drug abuse within the past 2 years prior to screening.
* Women who are pregnant or lactating.
* Positive urine drug or alcohol results at screening or check-in.
* Positive urine cotinine at screening.
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
* Seated blood pressure is less than 90/40 mm Hg or greater than 140/90 mmHg at screening.
* Seated heart rate is lower than 40 beats per minute (bpm) or higher than 99 bpm at screening.
* Hemoglobin level below the lower limit of normal at screening.
* Have been on a diet incompatible with the on-study diet, in the opinion of the PI, within the 28 days prior to the first dose of study drug, and throughout the study.
* Unable to refrain from or anticipates the use of any protocol defined drugs.
* Donation of blood or significant blood loss within 56 days prior to the first dose of study drug.
* Plasma donation within 7 days prior to the first dose of study drug.

Part 1 Only:

* History or presence of clinically significant hypersensitivity or idiosyncratic reaction to ACP-196, calcium carbonate, related compounds, or any inactive ingredients.
* History or presence of liver disease.

Part 2 Only:

* History or presence of clinically significant hypersensitivity or idiosyncratic reaction to ACP-196, omeprazole, related compounds or any inactive ingredients.
* History or presence of liver disease; Clostridium difficile-associated diarrhea.

Part 3 Only:

* History or presence of clinically significant hypersensitivity or idiosyncratic reaction to ACP-196, rifampin, related compounds, or any inactive ingredients.
* History or presence of liver disease; diabetes mellitus.
* Estimated creatinine clearance < 90 mL/min at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-09-21 (Actual); Primary Completion 2014-10-16 (Actual); Study Completion 2014-10-16 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of ACP-196 in Parts 1, 2, and 3 | Period 1: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for all parts; Period 2: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for Part 1, on Day 5 for Part 2, and on Days 1 and 9 for Part 3
Maximum Observed Plasma Concentration (Cmax) of ACP-196 in Parts 1, 2, and 3 | Period 1: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for all parts; Period 2: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for Part 1, on Day 5 for Part 2, and on Days 1 and 9 for Part 3

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time 0 to Time of Last Measurable Concentration (AUC0-last) of ACP-196 in Parts 1, 2, and 3 | Period 1: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for all parts; Period 2: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for Part 1, on Day 5 for Part 2, and on Days 1 and 9 for Part 3
Percent of AUC0inf Extrapolated (AUC%extrap) of ACP-196 in Parts 1, 2, and 3 | Period 1: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for all parts; Period 2: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for Part 1, on Day 5 for Part 2, and on Days 1 and 9 for Part 3
Area Under the Plasma Concentration-time Curve From Time 0 to 24 hours (AUC0-24h) of ACP-196 in Parts 1, 2, and 3 | Period 1: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for all parts; Period 2: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for Part 1, on Day 5 for Part 2, and on Days 1 and 9 for Part 3
Time to Reach Maximum Observed Plasma Concentration (Tmax) of ACP-196 in Parts 1, 2, and 3 | Period 1: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for all parts; Period 2: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for Part 1, on Day 5 for Part 2, and on Days 1 and 9 for Part 3
Apparent Terminal Elimination Half-life (T1/2) of ACP-196 in Parts 1, 2, and 3 | Period 1: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for all parts; Period 2: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for Part 1, on Day 5 for Part 2, and on Days 1 and 9 for Part 3
Apparent Terminal Elimination Rate Constant (λz) of ACP-196 in Parts 1, 2, and 3 | Period 1: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for all parts; Period 2: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for Part 1, on Day 5 for Part 2, and on Days 1 and 9 for Part 3
Apparent Total Body Clearance (CL/F) of ACP-196 in Parts 1, 2, and 3 | Period 1: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for all parts; Period 2: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 hrs on Day 1 for Part 1, on Day 5 for Part 2, and on Days 1 and 9 for Part 3
Incidence of Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events in Parts 1, 2, and 3 | From Day 1 through 14 days after the last dose (approximately 1 month) in all 3 parts
Number of Participants With Abnormal Physical Examinations and Vital Signs Reported as TEAEs in Parts 1, 2, and 3 | Part 1: Day 1; Part 2: Day 1 through Day 5; Part 3: Day 1 through Day 9
Number of Participants With Abnormal Electrocardiograms (ECGs) Reported as TEAEs in Parts 1, 2, and 3 | Part 1: Day 1; Part 2: Day 1 through Day 5; Part 3: Day 1 through Day 9
Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs in Parts 1, 2, and 3 | Part 1: Day 1; Part 2: Day 1 through Day 5; Part 3: Day 1 through Day 9

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hamdy, MD, Study Director — Acerta Pharma BV
Locations (1):
- Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home